CLINICAL TRIAL: NCT06115304
Title: Postprandial Profiles of Metabolites and Appetite-regulating Hormones in Plasma and Cerebrospinal Fluid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mikkel Bring Christensen (Other)
Responsible Party: Sponsor-Investigator, Mikkel Bring Christensen, Chief consultent at the department of Clinical Pharmacology, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CSF-meal
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Other)
  Interventions: Other: Large liquid meal, spinal catheter and venous line

INTERVENTIONS:
Other: Large liquid meal, spinal catheter and venous line — Large liquid meal (e.g. Nutricia® Energy 500 ml (750 kcal) admixed paracetamol 1000 mg (for estimation of gastric emptying).
  Spinal catheter for 4 hours, with samples taken at one hour interval.
  2 venous lines, one for saline and one for venous sampling every half hour

SUMMARY:
Overweight and obesity are rising in prevalence and becoming a growing threat to public health. Obesity is associated with an increased all-cause mortality, impaired quality of life, and numerous of disorders. Therapeutic strategies against obesity - which include an abundance of dietary and physical training programmes and pharmaceutical drugs to increase energy expenditure or limit appetite or gastro-intestinal fat absorption - have shown limited success on long term weight loss. Thus, overweight and associated conditions is becoming the new normal and there is a need for better understanding gut-to-brain signalling, hormonal and metabolic disturbances in overweight individuals.

The purpose of this health science research project is to describe the coinciding plasma and cerebrospinal fluid (CSF) profiles of selected biomarkers after co-ingestion of a meal and model pharmaceuticals in patients with overweight and/or type 2 diabetes compared to healthy control individuals.

ELIGIBILITY:
Inclusion Criteria:

* 10 male patients with obesity (BMI >30) and type 2 diabetes
* 10 male volunteers with normal weight (BMI 20-24) matched by age
* 10 male volunteers with obesity (BMI >30) matched by age

Exclusion Criteria:

1. Unwillingness to participate or wish to withdraw from ongoing protocol
2. Hepatic disease or hemorrhagic diatheses (including abnormal International Normalized Ratio (INR), bilirubin, blood levels of thrombocytes, alanine-aminotransferase (ALAT))
3. Anticoagulant treatment (e.g. treatment with warfarin, apixaban or another oral anticoagulant)
4. Anaemia (p-hemoglobin below normal range)
5. Nephropathy (se-creatinine >130 μM and/or albuminuria)
6. Suspected difficult access to the spinal canal (e.g. pronounced scoliosis, spinal stenosis, osteoporotic coincidence in the lower back, spina bifida, meningocele after surgical intervention)
7. Lumbar skin infection (e.g. herpes zoster, pustules or ulcers)
8. Medical history with headaches - both in connection with dura puncture and frequent headaches of other types
9. Central nervous system disease (including dementia, previous stroke, multiple sclerosis, epilepsy, etc.)
10. Clinical suspicion of increased intracranial pressure (headaches, visual disturbances etc.)
11. Patients with type 2 diabetes: Treatment with DPP-4 inhibitor or GLP-1 receptor agonist. Late diabetic complications including proliferative diabetic retinopathy (anamnestic), arteriosclerotic cardiovascular disease (heart failure or previous ischemic event/myocardial infarction)

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-10-05 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Appetite regulating hormones measured by specific immunoassays | After 1 hour
Appetite regulating hormones measured by specific immunoassays | After 2 hour
Appetite regulating hormones measured by specific immunoassays | After 3 hours
Appetite regulating hormones measured by specific immunoassays | After 4 hours

OTHER OUTCOMES:
Metabolomics measured in blood and cerebrospinalfluid using mass spectrometry | After 1 hour
Metabolomics measured in blood and cerebrospinalfluid using mass spectrometry | After 2 hours
Metabolomics measured in blood and cerebrospinalfluid using mass spectrometry | After 3 hours
Metabolomics measured in blood and cerebrospinalfluid using mass spectrometry | After 4 hours
Proteomics measured in blood and cerebrospinalfluid using mass spectrometry | After 1 hour
Proteomics measured in blood and cerebrospinalfluid using mass spectrometry | After 2 hours
Proteomics measured in blood and cerebrospinalfluid using mass spectrometry | After 3 hours
Proteomics measured in blood and cerebrospinalfluid using mass spectrometry | After 4 hours
Peptidomics measured in blood and cerebrospinalfluid using mass spectrometry | After 1 hour
Peptidomics measured in blood and cerebrospinalfluid using mass spectrometry | After 2 hour
Peptidomics measured in blood and cerebrospinalfluid using mass spectrometry | After 3 hours
Peptidomicsmeasured in blood and cerebrospinalfluid using mass spectrometry | After 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel.bring.christensen@regionh.dk B Christensen, MD, PhD, Principal Investigator — Department of clinical pharmacology, Bispebjerg Hospital
Locations (1):
- Deparrtment of clinical pharmacology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No